CLINICAL TRIAL: NCT02177786
Title: A Phase 2, Double-Blind, Placebo-Controlled, Dose-Ranging Study Evaluating the Efficacy, Safety, and Tolerability of GS-4997 in Subjects With Diabetic Kidney Disease
Brief Title: Efficacy, Safety, and Tolerability of Selonsertib (GS-4997) in Participants With Diabetic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-223-1015
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Gilead
MeSH Terms: conditions — Diabetic Nephropathies | interventions — selonsertib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Selonsertib 2 mg (Experimental): Participants will receive selonsertib 2 mg for 48 weeks.
  Interventions: Drug: Selonsertib
- Selonsertib 6 mg (Experimental): Participants will receive selonsertib 6 mg for 48 weeks.
  Interventions: Drug: Selonsertib
- Selonsertib 18 mg (Experimental): Participants will receive selonsertib 18 mg for 48 weeks.
  Interventions: Drug: Selonsertib
- Placebo to match selonsertib (Placebo Comparator): Participants will receive placebo to match selonsertib for 48 weeks.
  Interventions: Drug: Placebo to match selonsertib

INTERVENTIONS:
Drug: Selonsertib — Tablets administered orally once daily
  Other Names: GS-4997
  Arms: Selonsertib 18 mg; Selonsertib 2 mg; Selonsertib 6 mg
Drug: Placebo to match selonsertib — Tablets administered orally once daily
  Arms: Placebo to match selonsertib

SUMMARY:
The primary objective of this study is to determine the effect of selonsertib (formerly GS-4997) on estimated glomerular filtration rate (eGFR) decline in participants with diabetic kidney disease (DKD). Participants will be randomized with a 1:1:1:1 allocation to receive 1 of 3 doses of selonsertib (2 mg, 6 mg, or 18 mg) or matching placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult male or females with prior diagnosis of Diabetic Kidney Disease
* Type 2 diabetes mellitus diagnosis for at least 6 months
* eGFR (MDRD) at screening ≥ 15 mL/min/1.73m^2 to < 60 mL/min/1.73m^2
* Urine albumin to creatinine ratio (UACR) as follows:

  * Stage/Stratum 3a: eGFR range 45 to < 60 mL/min; UACR ≥ 600 mg/g
  * Stage/Stratum 3b: eGFR range 30 to < 45 mL/min; UACR ≥ 300 mg/g
  * Stage/Stratum 4: eGFR range 15 to < 30 mL/min; UACR ≥ 150 mg/g
* Receiving angiotensin-converting-enzyme inhibitor (ACEi) or angiotensin receptor blockers (ARB) at a minimum dose deemed appropriate for the individual by the investigator and be at a stable dose for the last three months

  * Individuals not on ACEi/ARB may be screened if there is documented intolerance to ACE inhibitor and/or ARB

Key Exclusion Criteria:

* Type 1 diabetes mellitus
* HbA1c > 9.5%
* Non-diabetic kidney disease
* UACR > 5000 mg/g on any measurement during screening
* End stage renal disease (ESRD; receiving peritoneal dialysis, hemodialysis, or status post renal transplantation) or anticipated to occur within the treatment period
* Unstable cardiovascular disease
* Pregnant or lactating females

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (104):
- United States (99):
  - The University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Chase Medcare, Huntsville, Alabama
  - Choice Medicine, Toney, Alabama
  - Akdhc Medical Research Services, Llc, Peoria, Arizona
  - Akdhc Medical Research Services, Llc, Phoenix, Arizona
  - Akdhc Medical Research Services, Llc, Prescott, Arizona
  - Robert J. Bloomberg, MD, Tempe, Arizona
  - AKDHC East Office, Tucson, Arizona
  - Clinical Research Connections, LLC, Harrisburg, Arkansas
  - North America Research Institute, Azusa, California
  - California Institute of Renal Research, Chula Vista, California
  - California Institute of Renal Research Inc., El Centro, California
  - Renal Consultants Medical Group Granada Hills, Granada Hills, California
  - Torrance Clinical Research, Lomita, California
  - IMD Medical Group, Los Angeles, California
  - Academic Medical Research Institute, Los Angeles, California
  - Kidney Research Center, Lynwood, California
  - Apex Research of Riverside, Riverside, California
  - San Francisco General Hospital, San Francisco, California
  - Clearview Medical Research, LLC, Santa Clarita, California
  - American Institute of Research, Whittier, California
  - Omega Research Consultants, DeBary, Florida
  - Creekside Medical Research, DeLand, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - ASA Clinical Research, Jupiter, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - The Chappel Group LLC, Kissimmee, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Prestige Clinical Research Center Inc, Miami, Florida
  - International Physicians Research / Nephrology Associates of South Miami, Miami, Florida
  - Tellus Clinical Research, Inc, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Central Florida Internists, Orlando, Florida
  - Sunset Point Medical Associates DBA, Palm Harbor, Florida
  - Pines Clinical Research Inc., Pembroke Pines, Florida
  - Central Florida Internists, Saint Cloud, Florida
  - Florida Pulmonary Research Institute, Winter Park, Florida
  - Rockdale Medical Research Associates, Conyers, Georgia
  - John H. Stroger Jr. Hospital Of Cook County, Chicago, Illinois
  - Midwest Endocrinology, Crystal Lake, Illinois
  - Beacon Medical Group Kidney and Hypertension Center, Mishawaka, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Hutchinson Clinic, P.A, Hutchinson, Kansas
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Research Nurse Specialists, LLc, Lafayette, Louisiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Internal Medicine Specialists, New Orleans, Louisiana
  - Green Clinic LLC, Ruston, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Southern Clinical Research, Zachary, Louisiana
  - Johns Hopkins Hospital/University, Baltimore, Maryland
  - A. Kaldun Nossuli MD Research, Bethesda, Maryland
  - Wayne State University, Detroit, Michigan
  - Apex Medical Research.Com, Flint, Michigan
  - Elite Clinical Research, Flint, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - VA Medical Center, Kansas City, Missouri
  - Mercury Street Medical Group, PLLC, Big Sky Clinical Research, LLC, Butte, Montana
  - Alegent Creighton Health, Omaha, Nebraska
  - Creighton Diabetes Center, Omaha, Nebraska
  - Nephrology and Hypertension Associates of New Jersey, Voorhees Township, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Nephrology Associates, PC, Flushing, New York
  - Mountain Kidney and Hypertension Associates, Asheville, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Carolina Research Center, Shelby, North Carolina
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Craig S Thompson MD LLC, Marion, Ohio
  - Your Diabetes Endocrine Nutrition Group Inc, Mentor, Ohio
  - Chris Sholer, MD, PC, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Knoxville Kidney Center, Knoxville, Tennessee
  - Arlington Nephrology, Arlington, Texas
  - MW Clinical Research Center, Beaumont, Texas
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Texas Tech Univ. Health Sciences Center, El Paso, Texas
  - TVC Clinical Research, Gonzales, Texas
  - Diagnostic Clinic of Houston, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Lakewood Family Practice, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - HMRI CCAT Pearland, Pearland, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Val R. Hansen, M.D., Bountiful, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Zablocki VAMC, Milwaukee, Wisconsin
- Canada (5):
  - BC Diabetes, Vancouver, British Columbia
  - Co-Medica Research Network, Courtice, Ontario
  - Clinical Research Solutions, Inc., Kitchener, Ontario
  - OTT Healthcare Inc., Scarborough Village, Ontario
  - Toronto East General Medical Centre, Toronto, Ontario

REFERENCES:
- [Result] Chertow GM, Pergola PE, Chen F, Kirby BJ, Sundy JS, Patel UD; GS-US-223-1015 Investigators. Effects of Selonsertib in Patients with Diabetic Kidney Disease. J Am Soc Nephrol. 2019 Oct;30(10):1980-1990. doi: 10.1681/ASN.2018121231. Epub 2019 Sep 10. PMID 31506292
- [Derived] Tesch GH, Ma FY, Han Y, Liles JT, Breckenridge DG, Nikolic-Paterson DJ. ASK1 Inhibitor Halts Progression of Diabetic Nephropathy in Nos3-Deficient Mice. Diabetes. 2015 Nov;64(11):3903-13. doi: 10.2337/db15-0384. Epub 2015 Jul 15. PMID 26180085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and Canada. The first participant was screened on 30 June 2014. The last study visit occurred on 22 August 2016.
Pre-assignment Details: 893 participants were screened.
Groups:
- Selonsertib 2 mg: Selonsertib 2 mg tablet once daily for 48 weeks
- Selonsertib 6 mg: Selonsertib 6 mg tablet once daily for 48 weeks
- Selonsertib 18 mg: Selonsertib 18 mg tablet once daily for 48 weeks
- Placebo: Placebo tablet once daily for 48 weeks
Period: Overall Study
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Started | 81 | 84 | 84 | 85
Randomized and Treated | 81 | 84 | 83 | 85
Completed | 75 | 70 | 66 | 72
Not Completed | 6 | 14 | 18 | 13
Not completed — Withdrew Consent | 2 | 6 | 9 | 5
Not completed — Progression to End Stage Renal Disease | 2 | 3 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 2 | 3
Not completed — Death | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0
Not completed — Missing study completion status | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo | Total
Number analyzed (Participants) | 81 | 84 | 83 | 85 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.1) | 62 (8.1) | 63 (9.0) | 62 (7.9) | 63 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 20 | 27 | 32 | 107
  Male | 53 | 64 | 56 | 53 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 31 | 33 | 30 | 119
  Not Hispanic or Latino | 56 | 53 | 50 | 55 | 214
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Race: Asian | 3 | 4 | 2 | 3 | 12
  Race: Black | 20 | 23 | 11 | 19 | 73
  Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1 | 0 | 2
  Race: White | 53 | 57 | 68 | 61 | 239
  Race: Other | 4 | 0 | 1 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 3 | 3 | 4 | 12
  United States | 79 | 81 | 80 | 81 | 321
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — The values of eGFR were calculated using the modification of diet in renal disease (MDRD) equation: eGFR = 175 x Serum Creatinine^-1.154 × age^-0.203 × 1.212 (if participant is black) × 0.742 (if female).
  mL/min/1.73 m^2 | 31.6 (10.92) | 31.9 (11.58) | 31.1 (10.44) | 31.4 (11.87) | 31.5 (11.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in eGFR From Baseline at Week 48
Description: The values of eGFR were calculated using the MDRD equation: eGFR = 175 x Serum Creatinine^-1.154 × age^-0.203 × 1.212 (if participant is black) × 0.742 (if female).
Time Frame: Baseline; Week 48
Population: Full Analysis Set included all randomized participants who took at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 81 | 84 | 83 | 85
mL/min/1.73 m^2 | -2.83 (0.86) | -2.37 (0.87) | -4.07 (0.89) | -3.20 (0.85)
Statistical Analysis 1: Comparison: Selonsertib 2 mg vs Placebo; Test type: Superiority; p = 0.755, MMRM — Data was calculated using a mixed-effect model repeated measures (MMRM) model including terms for treatment group, baseline eGFR, visit and treatment by visit interaction for comparison of change from baseline in eGFR between selonsertib and placebo; Least Square Means Difference = 0.38, 95% CI 2-sided [-2.00 to 2.75], Standard Error of Mean 1.21
Statistical Analysis 2: Comparison: Selonsertib 6 mg vs Placebo; Test type: Superiority; p = 0.492, MMRM — Data was calculated using a MMRM model including terms for treatment group, baseline eGFR, visit and treatment by visit interaction for comparison of change from baseline in eGFR between selonsertib and placebo; Least Square Means Difference = 0.84, 95% CI 2-sided [-1.55 to 3.23], Standard Error of Mean 1.22
Statistical Analysis 3: Comparison: Selonsertib 18 mg vs Placebo; Test type: Superiority; p = 0.481, MMRM — [p-value comment as in outcome 1, analysis 2]; Least Square Means Difference = -0.87, 95% CI 2-sided [-3.29 to 1.56], Standard Error of Mean 1.23

2. Secondary Outcome: Percentage of Participants Achieving at Least a 30% Reduction From Baseline in Albuminuria (As Measured by Urine Albumin to Creatinine Ratio) at Week 48
Description: Baseline was the average of the last 2 values prior to randomization and the last value on or after the randomization date, but prior to or on the first dose date. Urine Albumin to Creatinine Ratio= urine albumin/urine creatinine.
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Number analyzed (Participants) | 81 | 84 | 83 | 85
percentage of participants | 28.4 | 21.4 | 27.7 | 30.6
Statistical Analysis 1: Comparison: Selonsertib 2 mg vs Placebo; Test type: Superiority; p = 0.798, Cochran-Mantel-Haenszel; P-value was based on a Cochran-Mantel-Haenszel (CMH) test stratified by stage of disease to compare the response rate between selonsertib and placebo; Difference in Percentages = -2.2, 95% CI 2-sided [-16.1 to 11.7] — The 95% confidence interval (CI) in the difference in percentages between selonsertib and placebo was based on Wald Asymptotic test
Statistical Analysis 2: Comparison: Selonsertib 6 mg vs Placebo; Test type: Superiority; p = 0.175, Cochran-Mantel-Haenszel; P-value was based on a CMH test stratified by stage of disease to compare the response rate between selonsertib and placebo; Difference in Percentages = -9.2, 95% CI 2-sided [-22.3 to 4.0] — The 95% CI in the difference in percentages between selonsertib and placebo was based on Wald Asymptotic test
Statistical Analysis 3: Comparison: Selonsertib 18 mg vs Placebo; Test type: Superiority; p = 0.686, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 2]; Difference in Percentages = -2.9, 95% CI 2-sided [-16.6 to 10.9] — The 95% CI in the difference in percentages between selonsertib and placebo was based on Wald Asymptotic test

ADVERSE EVENTS:
Time Frame: First dose date up to Week 48 plus 30 days
Description: Safety Analysis Set included all randomized participants who took at least 1 dose of study drug.
Arm/Group | Selonsertib 2 mg | Selonsertib 6 mg | Selonsertib 18 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 24/81 | 20/84 | 20/83 | 16/85
Other Adverse Events (participants affected / at risk) | 51/81 | 47/84 | 55/83 | 48/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib 2 mg (N=81) | Selonsertib 6 mg (N=84) | Selonsertib 18 mg (N=83) | Placebo (N=85)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 4 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Electrocardiogram ST segment abnormal (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 1 | 2
Bladder mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selonsertib 2 mg (N=81) | Selonsertib 6 mg (N=84) | Selonsertib 18 mg (N=83) | Placebo (N=85)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 7 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 7 | 4
Nausea (Gastrointestinal disorders) | 8 | 4 | 1 | 4
Oedema peripheral (General disorders) | 2 | 5 | 4 | 7
Bronchitis (Infections and infestations) | 1 | 1 | 3 | 5
Cellulitis (Infections and infestations) | 1 | 3 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 8 | 8
Urinary tract infection (Infections and infestations) | 5 | 1 | 5 | 4
Blood creatinine increased (Investigations) | 6 | 1 | 3 | 2
Gout (Metabolism and nutrition disorders) | 3 | 5 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3 | 7 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 4 | 4 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 6 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 5 | 4
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 5 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 5 | 3 | 3
End stage renal disease (Renal and urinary disorders) | 2 | 3 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 3
Hypertension (Vascular disorders) | 7 | 6 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years